CLINICAL TRIAL: NCT03766139
Title: Evaluation of Supercell Glue (Platelet Rich Fibrin Matrix{PRFM} AND Peripheral Blood Mesenchymal Stem Cells {PBMSCs} ) as a Regenerative Material in Human Mandibular Periodontal Intraosseous Defect - A Split Mouth Randomized Controlled Trial
Brief Title: Regenerative Potential of Supercell Glue and Platelet Rich Fibrin Matrix
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KLE Society's Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr Laveena Singhal, Principal investigator, KLE Society's Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PARVATHY61
Record Dates: First submitted 2018-08-13; First posted 2018-12-06 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Intrabony Periodontal Defect

STUDY DESIGN:
Intervention Model Description: The study will be a Double Blinded Randomized controlled clinical trial with a split mouth design.
Who Masked: Participant, Investigator
Masking Description: The sites will be randomly (computer generated tabulation method) assigned into control group (treated with PRFM alone) and test group (treated with Supercell Glue).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SUPERCELL GLUE(STEM CELLS AND PRFM) (Experimental): Following optimum anaesthesia, reflection of full thickness mucoperiosteal flaps for defect access and thorough debridement will be done. Subsequently the defect will be filled with supercell glue in test sites .
  Interventions: Biological: SUPERCELL GLUE
- PRFM ALONE (Active Comparator): Following optimum anaesthesia, reflection of full thickness mucoperiosteal flaps for defect access and thorough debridement will be done. Subsequently the defect will be filled with PRFM in control sites
  Interventions: Biological: PRFM ALONE

INTERVENTIONS:
Biological: SUPERCELL GLUE — Following optimum anaesthesia, reflection of full thickness mucoperiosteal flaps for defect access and thorough debridement will be done. Subsequently the defect will be filled with supercell glue in test sites (randomly selected by computer generated tabulation method)
  Arms: SUPERCELL GLUE(STEM CELLS AND PRFM)
Biological: PRFM ALONE — Following optimum anaesthesia, reflection of full thickness mucoperiosteal flaps for defect access and thorough debridement will be done. Subsequently the defect will be filled with PRFM in control sites(randomly selected by computer generated tabulation method)
  Arms: PRFM ALONE

SUMMARY:
Utilizing the osteogenic properties of both platelet rich fibrin matrix and peripheral blood mesenchymal stem cells for periodontal regeneration would be novel and may be advantageous than using Platelet rich fibrin matrix alone. The literature search does not show any human clinical trial conducted till date to assess the regenerative potential of this new material i.e. Supercell glue (PRFM and PBMSCs).In this new material because of the addition of a patented gel the second spin to procure the PRFM has been eliminated and this seems to be an additional advantage. This study therefore aims at the evaluation of Supercell glue (PRFM and PBMSCs) as a regenerative material in comparison with PRFM alone in human mandibular periodontal intraosseous defects.

DETAILED DESCRIPTION:
Periodontal regeneration involves the formation of alveolar bone, cementum and a new functional periodontal ligament. Over the recent years the concept of periodontal treatment has focused towards regeneration with a goal of regaining natural periodontal apparatus. Numerous procedures have been investigated in the past to try to promote periodontal regeneration which range from root biomodifications, soft tissue grafts, bone replacement grafts, guided tissue regeneration to the use of combinations of the same. However the success of these approaches are highly variable. As a consequence current research trends are inclined towards the principle of 'biological solutions for biological problem' and thus attempts are directed towards various approaches like tissue engineering, ERT (endogenous regenerative technology), application of biologics, cell based techniques, biomimetic nanoscaffold fabrication and others for periodontal regeneration. Of all known Polypeptide Growth Factors, Platelet Derived Growth Factor (PDGF) and Transforming Growth Factor β (TGF β) which are abundant in α granule of platelets are shown to exert a favourable effect on periodontal regeneration. Therefore use of platelet concentrates is a convenient approach to obtain autologous growth factors.

Platelet rich fibrin matrix (PRFM) is an autologous concentrated platelet-rich thrombin free fibrin matrix, prepared by two step centrifugation of blood. Platelets isolated, remain intact and retain their growth factor compliment. This allows a more effective, sustained release of growth factors to the wound site following PRFM application. During the second spin, a cross-linking of fibrin takes place, resulting in the formation of a dense fibrin matrix, within which a concentration of viable platelets can be found. Having an organized fibrin matrix at the start of healing accelerates the speed of vascular ingress into the wound compared to non-accelerated healing, which requires a longer time for fibrin formation and the development of vascularity. The earlier the vascularity is established, faster is the migration of the bone-forming cells at the wound site and initiation of bone formation. Therapeutic applications of platelet-rich products have led to improved bone regeneration.

Mesenchymal stem cells (MSCs) are a multipotent stromal cells with prominent regenerative functions. MSCs were first identified and isolated from bone marrow and then found in various tissues including umbilical cord, adipose tissue and peripheral blood. Among these sources peripheral blood MSCs draw increasing attention as they share similar biological characteristics with MSCs derived from bone marrow or adipose tissue. Bone marrow derived mesenchymal stem cells(BMMSCs) are multipotent cells capable of differentiating into osteoblasts, chondrocytes, adipocytes, fibroblasts, tenocytes, and myoblasts, which are considered as a cell source for various tissue repair and regenerating bone defects. The requirements of aspiration of bone marrow from the patient will cause pain and morbidity of the donor sites. It will be very convenient if peripheral blood mesenchymal stem cells (PBMSCs) could be harvested and expanded to enough numbers, with their osteogenic capacity maintained in a clinical permitted period.

Hence, utilizing the osteogenic properties of both platelet rich fibrin matrix and peripheral blood mesenchymal stem cells for periodontal regeneration would be novel and may be advantageous than using Platelet rich fibrin matrix alone. The literature search does not show any human clinical trial conducted till date to assess the regenerative potential of this new material i.e. Supercell glue (PRFM and PBMSCs).In this new material because of the addition of a patented gel the second spin to procure the PRFM has been eliminated and this seems to be an additional advantage. This study therefore aims at the evaluation of Supercell glue (PRFM and PBMSCs) as a regenerative material in comparison with PRFM alone in human mandibular periodontal intraosseous defects.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients diagnosed with chronic periodontitis.
* Patients with mandibular infrabony pocket measuring ≥ 6mm with radiographic evidence of intrabony defect

Exclusion Criteria:

* Pregnant /lactating women
* Patients taking any drug known to affect the number and function of platelets in the past 3 months.
* Patients with abnormal platelet count.
* Patients with immunologic diseases
* Current smokers.
* History of periodontal therapy in the last 6 months.
* Any other contraindications for periodontal surgery.
* Maxillary intrabony defect.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Early wound healing index (Supercell in early wound healing index) | 1 week
  early wound healing index in intraosseous periodontal defects
Change in probing pocket depth and clinical attachment gain (Supercell as a regenerative novel material) | baseline,3 months,6 months
  Change in probing pocket depth reduction and clinical attachment gain measured in millimetres in intraosseous defects
Change in the bone level (Supercell as a biological material) | baseline, 3 months,6 months
  change in the bone level will be assessed radiographically using Image J analysis software measured in millimeters
Change in the clinical parameters of gingival index and plaque index (Supercell as a regenerative material using clinical indices) | baseline,3 months,6 months
  change in the clinical parameters of gingival index and plaque index (no units as these are indices) in intraosseous periodontal defects

CONTACTS AND LOCATIONS:
Locations (1):
- Kle Society'S Institute of Dental Sciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided